CLINICAL TRIAL: NCT04608357
Title: Integrated Patient Avatars for Guiding Systemic Therapy Treatments: "Intuition-Free" Decisions in Metastatic Breast Cancer Patients
Brief Title: Integrated Patient Avatars for Guiding Systemic Therapy Treatments in Metastatic Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: AFP Innovation Fund (Other)
Responsible Party: Principal Investigator, Dr. Katarzyna Jerzak, Medical Oncologist & Associate Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: SUN-2252
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Breast Neoplasms; Metastatic Breast Cancer; Cancer, Breast
Keywords: metastatic breast cancer; systemic therapy; needle core biopsy; PDXovo; feasibility study; tumor take rate
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Large-Core Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — needle core biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Needle Core Biopsies — Not an interventional study

SUMMARY:
The investigators propose to use clinically validated patient avatar technology ("PDXovo") that can test multiple drugs against patients' cancers to identify the most promising systemic therapy for each individual.

DETAILED DESCRIPTION:
The primary goal of this feasibility study is to determine the percentage of patients for whom PDXs are successfully generated within 7-10 days. This will give the investigators an indication of the success rate for providing patients with actionable information if this PDX technology were to be implemented in the clinic. Since the PDXs will also receive the same drug as the patient, there is an opportunity to assess the agreement between the clinical response and the PDX response.

As a secondary goal, the response of PDXs will be compared to the patient's response to systemic therapy, as measured using the objective response rate at 12 weeks +/- 4 weeks (ORR, measured using RECIST 1.1 criteria).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+.
2. Metastatic breast cancer irrespective of subtype.
3. Measurable disease as per RECIST 1.1 criteria.
4. Metastatic disease involving the lymph nodes and/or visceral organs is required.
5. Willingness to undergo a biopsy prior to the start of planned systemic therapy.

Exclusion Criteria:

1. Lack of feasibility to obtain a core biopsy of a metastatic site other than the bone (e.g. a metastatic lesion cannot be safely sampled due to proximity to vasculature).
2. Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic breast cancer irrespective of subtype prior to receiving either front-line or subsequent line systemic therapy
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determine the tumor take rate in PDX | 7-10 days
  perform a feasibility study to determine the tumor take rate(s) in PDXs generated from needle core biopsies collected from metastatic breast cancer patients

SECONDARY OUTCOMES:
Compare response rates of PDXs & with that of the patient from whom the PDX was derived | 8 to 16 weeks
  The response of PDXs will be compared to the patient's response to systemic therapy, as measured using the objective response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna J Jerzak, MD MSc FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grafinger OR, Hayward JJ, Meng Y, Geddes-McAlister J, Li Y, Mar S, Sheng M, Su B, Thillainadesan G, Lipsman N, Coppolino MG, Trant JF, Jerzak KJ, Leong HS. Cancer cell extravasation requires iplectin-mediated delivery of MT1-MMP at invadopodia. Br J Cancer. 2024 Sep;131(5):931-943. doi: 10.1038/s41416-024-02782-9. Epub 2024 Jul 5. PMID 38969866